CLINICAL TRIAL: NCT00092118
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study Investigating the Clinical Effects of Montelukast in Patients With Perennial Allergic Rhinitis
Brief Title: The Clinical Effects of Montelukast in Patients With Perennial Allergic Rhinitis (0476-265)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-265; MK0476-265; 2004_018
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Results first posted 2010-07-23 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Montelukast
  Interventions: Drug: Montelukast
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Montelukast — one 10 mg tablet, taken once daily at bed time for 6 weeks
  Arms: 1
Drug: Comparator: Placebo — one placebo tablet, taken once daily at bed time for 6 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of an approved medication on the symptoms of perennial allergic rhinitis (an inflammation of the mucous membrane of the nose similar to that found in hay fever except that symptoms persist throughout the year), in patients who have a history of perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker with a 2-year documented history of perennial allergic (symptoms that persist throughout the year) rhinitis symptoms and positive allergy testing

Exclusion Criteria:

* Medical history of a lung disorder (other than asthma) or a recent upper respiratory tract infection

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1992 (Actual)
Dates: Start 2003-10; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Patel P, Philip G, Yang W, Call R, Horak F, LaForce C, Gilles L, Garrett GC, Dass SB, Knorr BA, Reiss TF. Randomized, double-blind, placebo-controlled study of montelukast for treating perennial allergic rhinitis. Ann Allergy Asthma Immunol. 2005 Dec;95(6):551-7. doi: 10.1016/S1081-1206(10)61018-6. PMID 16400895

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened at 122 sites worldwide.
  Primary therapy period: Oct 2003 to May 2004
Pre-assignment Details: Patients who required excluded medication and those who did not meet a minimum predefined level of combined daytime nasal symptoms score during the run-in period were excluded from randomization.
Groups:
- Placebo: Montelukast matching-image placebo tablets were taken orally once daily at bedtime for 6 weeks.
- Montelukast 10 mg: Montelukast 10 mg tablets were taken orally once daily at bedtime for 6 weeks.
Period: Overall Study
Arm/Group | Placebo | Montelukast 10 mg
Started | 990 (1 patient discontinued after randomization due to a adverse experience that began pre-randomization.) | 1002 (2 patients discontinued after randomization due to adverse experience that began pre-randomization.)
Completed | 906 | 913
Not Completed | 84 | 89
Not completed — Adverse Event | 35 | 32
Not completed — Lack of Efficacy | 12 | 14
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 23 | 25
Not completed — Withdrawal by Subject | 4 | 10
Not completed — Other | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Montelukast 10 mg | Total
Number analyzed (Participants) | 990 | 1002 | 1992
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (13.12) | 36.3 (13.61) | 36.4 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 632 | 644 | 1276
  Male | 358 | 358 | 716
Daytime nasal symptoms score [Mean (Standard Deviation); unit: Scores on a scale] — Computed using the average values of the 3 individual daytime nasal symptoms scores of congestion, rhinorrhea, and sneezing on a 4-point scale [Score 0 (best) to 3 (worst)]. Baseline is computed as the average daily value during the prerandomization run-in period (which included the 5-7 days prior to randomization at Visit 3).
  Scores on a scale | 2.10 (0.41) | 2.09 (0.40) | 2.10 (0.41)
Rhinoconjunctivitis Quality-of-Life Score [Mean (Standard Deviation); unit: Score on a scale] — Patients completed the validated, self-administered RQLQ which
  included 28 items on a 7-point scale [Score 0 (best) to 6 (worst)] across 7 domains: activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional. The scores within each domain were averaged, then the scores for the 7 domains were averaged to obtain the overall score. Baseline is the Visit 3 value.
  Score on a scale | 2.96 (1.10) | 2.94 (1.04) | 2.95 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daytime Nasal Symptoms Score Averaged Over the 6-week Treatment Period in Patients With Perennial Allergic Rhinitis
Description: Mean change from baseline in Daytime Nasal Symptoms score averaged over the 6-week treatment period. The Daytime Nasal Symptoms score was calculated as the average of the 3 individual scores for Congestion, Rhinorrhea, and Sneezing, each rated by patients daily on a 4-point scale [Score 0 (best) to 3 (worst)].
Time Frame: 6 week treatment period (from baseline though the end of week 6)
Population: The primary efficacy analyses were performed using a modified intention-to-treat (MITT) approach. All patients with efficacy measurements, both at baseline and during the treatment period were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 980 | 1000
Score on a scale | -0.37 [-0.40 to -0.34] | -0.44 [-0.48 to -0.41]

2. Secondary Outcome: Patient's Global Evaluation of Allergic Rhinitis at the End of the 6 Week Treatment Period
Description: An evaluation by the patient, administered at the last visit (or upon discontinuation) using a 7-point scale [Score 0 (best) to 6 (worst)], in answer to a single question regarding the change in symptoms as compared to the beginning of the study.
Time Frame: At the end of the 6 week treatment period
Population: The analysis was performed using a modified intention-to-treat (MITT) approach. Patients were excluded if no treatment period data were available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 969 | 977
Score on a scale | 2.42 [2.33 to 2.51] | 2.27 [2.18 to 2.35]

3. Secondary Outcome: Mean Change From Baseline in Rhinoconjunctivitis Quality-of-life Questionnaire (RQLQ) Overall Score After the 6 Week Treatment Period
Description: Patients completed the validated, self-administered RQLQ which included 28 items on a 7-point scale [Score 0 (best) to 6 (worst)] across 7 domains: activities, sleep, nonnose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional. The scores for each domain were averaged, then scores for the 7 domains were averaged to obtain the overall score.
Time Frame: Baseline and Week 6
Population: The primary efficacy analyses were performed using a modified intention-to-treat (MITT) approach. Patients were excluded if no baseline or treatment period data were available
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 969 | 977
Score on a scale | -0.69 [-0.76 to -0.62] | -0.84 [-0.91 to -0.77]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected during the 6 week, double-blind treatment period, and up to and including 14 days after the last dose of study therapy.
Description: The number of participants listed in the AE tables (990 placebo & 1002 montelukast) is the number that received treatment.
  Although a participant may have 2 or more AEs they are counted only once in a category. The same participant may appear in other categories.
Arm/Group | Placebo | Montelukast 10 mg
Serious Adverse Events (participants affected / at risk) | 1/990 | 4/1002
Other Adverse Events (participants affected / at risk) | 0/990 | 0/1002
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=990) | Montelukast 10 mg (N=1002)
Myocardial Infarction (Cardiac disorders) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Anxiety Disorder (Psychiatric disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.